CLINICAL TRIAL: NCT06695546
Title: Evaluation of the Venous Excess Ultrasound Score (VExUS) After Circulating Volume Modification in Children. VExUS-Mod
Brief Title: Evaluation of the Venous Excess Ultrasound Score (VExUS) After Circulating Volume Modification in Children.
Acronym: VExUS-Mod
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0457
Record Dates: First submitted 2024-11-08; First posted 2024-11-19 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Blood Volume Expansion
Keywords: extra renal purification; bleeding; vascular filling
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients over one year of age treated at Toulouse University Hospital and receiving extrarenal purification, bloodletting or vascular filling > 10 ml/kg.
  Interventions: Other: VExUS evaluation ultrasound

INTERVENTIONS:
Other: VExUS evaluation ultrasound — VExUS evaluation by ultrasound will be performed before the filling/bleeding/cleaning procedure, and again after the procedure:
  * Inferior vena cava measurement in Time-Motion (TM) mode, 1-2 cm from the right atrial orifice.
  * Hepatic venous Doppler measurement in pulsed Doppler mode.
  * Renal vein Doppler measurement in pulsed Doppler mode. Each measurement is performed three times consecutively (to average the results), then the ultrasound measurements are compiled into a score according to the degree of doppler severity.

SUMMARY:
Venous overload has an impact on peripheral organ perfusion and on the short- and long-term prognosis of intensive care patients. The VExUS ultrasound score is a new tool whose parameters can be used to estimate this impact. This score was initially evaluated and validated on an adult population. ) In children, there is only one study looking at the use and applicability of this VExUS score, highlighting its feasibility in a paediatric population, as well as a possible correlation between elevated central venous pressure and altered renal Doppler (one of the score's components).

ELIGIBILITY:
Inclusion Criteria:

Children aged between 1 and 18 years, receiving extrarenal purification with UF > 10 ml/kg, bleeding > 10 ml/kg or vascular filling > 10 ml/kg

Exclusion Criteria:

* Refusal of the patient or opposition of one or both holders of parental authority.
* Minors with parental authority.
* Ultrafiltration time > 6h.
* Curarized patient, known abnormality of the hepatorenal venous network.
* Patient agitated or poor tolerance of the examination.
* Parents under court protection, guardianship or curatorship.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children aged between 1 and 18 years, receiving extrarenal purification with UF > 10 ml/kg, bleeding > 10 ml/kg or vascular filling > 10 ml/kg treated at Toulouse University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Change in VExUS score | 10 minutes before en after the procedure of extrarenal purification, bloodletting or vascular filling
  The correlation between ultrasound measurement of the VExUS score and the change in blood volume induced by extrarenal purification, bloodletting or vascular filling is studied. Ultrasound is performed before and after the procedure, each measure 3 times in succession, to establish the score.

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat SIERRA COLOMINA, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No